CLINICAL TRIAL: NCT02123563
Title: Evaluation of Mechanical-chemical Gingival Therapy in Diabetic, Obese or Diabese Subjects: Quantitative and Qualitative Analysis of Local and General Aspects.
Brief Title: Mechanical-chemical Gingival Therapy in Diabetics and/or Obese
Acronym: MCGTDO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Taubate (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010/20424-1; 522/10 (Other: Ethics Committee Approval)
Record Dates: First submitted 2014-04-09; First posted 2014-04-25 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Gingivitis; Diabetes; Obesity
MeSH Terms: conditions — Gingivitis; Diabetes Mellitus; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrason Essential oils rinse (Experimental): Ultrasonic debridement followed by twice daily home use of an essential-oils mouth rinse (20mL, 30 seconds for each rinse) for 3 months
  Interventions: Other: Ultrason Essential oils rinse
- Ultrason Placebo rinse (Placebo Comparator): Ultrasonic debridement followed by twice daily home use of a placebo rinse (20mL, 30 seconds for each rinse) for 3 months
  Interventions: Other: Ultrason Placebo rinse

INTERVENTIONS:
Other: Ultrason Essential oils rinse — Test treatment strategy combined mechanical and chemical procedures. Mechanical procedures were: a) ultrasonic debridement to remove dental plaque, calculus and teeth staining; b) dental polishing and c) oral hygiene instructions related to brushing and flossing. Toothbrush, dental floss and fluoride dentifrice were monthly provided. Within the same visit participants performed at the study center the first supervised rinse. Other rinses were performed at home unsupervised. A diary card was used to register times of rinsing. Participants rinsed twice a day a commercially available non-prescription essential-oils solution (20mL, 30 seconds for each rinse) for 3 months. This solution is composed of eucalyptol 0.092%, menthol 0.042%, methyl salicylate 0.060%, thymol 0.064%, zinc chloride and sodium fluoride 0.0221%.
  Other Names: Listerine total care
  Arms: Ultrason Essential oils rinse
Other: Ultrason Placebo rinse — Comparative treatment strategy combined mechanical and chemical procedures. Mechanical procedures were: a) ultrasonic debridement to remove dental plaque, calculus and teeth staining; b) dental polishing and c) oral hygiene instructions related to brushing and flossing. Toothbrush, dental floss and fluoride dentifrice were monthly provided. Within the same visit participants performed at the study center the first supervised rinse. Other rinses were performed at home unsupervised. A diary card was used to register times of rinsing. Participants rinsed twice a day a placebo solution (20mL, 30 seconds for each rinse) for 3 months.
  Other Names: Placebo mouth rinse manipulated for the present study.
  Arms: Ultrason Placebo rinse

SUMMARY:
Diabetes and obesity affect many people in different countries. Similarly, millions of people have some type of gum disease such as gingivitis. The present study was conducted to clarify if systemic conditions such as diabetes and obesity could impair the response to gingivitis treatment. Subjects with gum disease showing diabetes type II (from 40 to 50 subjects), slight to moderate obesity (from 40 to 50 subjects) or its combination (from 40 to 50 subjects) were selected for the present study. In addition normal-weight subjects with gum disease (from 40 to 50 subjects) besides a group without gum disease (from 40 to 50 subjects) were selected for comparisons. After verbal and written explanations about the study, subjects who matched study criteria and who signed the informed consent form underwent full oral examinations in two separate visits. In the first visit, after a clinical examination to verify the levels of gingival inflammation and the accumulated amounts of dental plaque, the bone height was determined by X-Ray examinations. Bad breath was also evaluated by a chair-side apparatus. Additional laboratorial examinations included a) quantification of bacteria that cause gum disease from dental plaque samples, b) quantification of inflammatory products from gingival fluid sampling and c) quantification of produced saliva. Self-report questionnaires were used to check the impact of oral condition and treatment of gum disease in quality of life and individual daily performance. These examinations were repeated 3 months after dental treatment. All subjects received ultrasonic dental prophylaxis for cleaning their teeth. Based on systemic/oral conditions each group rinsed either an essential-oils containing mouth rinse or a placebo rinse. First rinse was supervised and the other ones were performed at home twice a day for three months. Each participant also received a toothbrush, a dental floss and a fluoride toothpaste monthly after oral hygiene instructions. Adherence to the treatment and occurrence of undesirable side effects were monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* plaque-related gingivitis (with no radiographic evidence of periodontal bone resorption and a bleeding site rate of more than 30%)
* periodontally healthy group (with no radiographic evidence of periodontal bone resorption and a bleeding site rate of less than 30%)
* at least 20 natural teeth
* diabetes group: controlled type II diabetes (with a blood glycated hemoglobin level between 6.5 and 7%) that was diagnosed at least 3 years but no more than 5 years prior to the study
* normal salivary flow
* obesity group: obesity level I - body mass index: 30 to 34.99 kg/m2 or obesity level II - body mass index: 35 to 39.99 kg/m2
* normal weight group: body mass index: 20 to 24.99 kg/m2;

Exclusion Criteria:

* gingival overgrowth
* orthodontic devices
* extended prosthetic fixed devices
* removable partial dentures or overhanging restorations
* systemic diseases or other conditions that could influence the periodontal status (other than diabetes within the diabetic group)
* overweight - BMI 25 to 29.99 kg/m2 and obesity level III or morbid obesity - ≥ 40 kg/m2 (obesity group) - alcohol abuse
* pregnancy or breast-feeding
* history of sensitivity or suspected allergies following the use of oral hygiene products
* the need for antibiotic prophylaxis; antibiotics and/or anti-inflammatory drug use in the six months prior to the beginning of the study
* regular use of chemotherapeutic antiplaque/antigingivitis products
* periodontal treatment performed within six months prior to study initiation
* unwillingness to return for follow-up

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 240 (Actual)
Dates: Start 2012-06; Primary Completion 2013-06 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
plaque and gingival indices | 3 months
  percentage of dental surfaces showing mild (scores 0,1), moderate (scores 2,3) or severe (scores 4,5) amounts of dental plaque or showing gingival bleeding (positive or negative) after gentle probing

CONTACTS AND LOCATIONS:
Locations (1):
- University of Taubate - Nucleus of periodontal research, Taubaté, São Paulo, Brazil